CLINICAL TRIAL: NCT05494151
Title: Investigation of the Metabolic Substrate of Patients With Myocardial Infarction and Derivation of a Risk Estimation Algorithm to Evaluate Cardiovascular Risk Beyond Standard Modifiable Risk Factors (SMuRFs) - (The MetaSMuRF Study)
Brief Title: Metabolic Substrate of Patients With Myocardial Infarction With and Without Modifiable Cardiovascular Risk Factors
Acronym: Meta-SMuRF
Status: Withdrawn | Type: Observational
Why Stopped: Due to unforeseen challenges in participant recruitment and retention, the study was early terminated to maintain the integrity of the data and ensure ethical standards were upheld.
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Dimitrios Moysidis, Cardiology Fellow, Aristotle University Of Thessaloniki
Other Study IDs: 64000/20-4-2022
Record Dates: First submitted 2022-08-06; First posted 2022-08-09 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Cardiovascular Diseases; Acute Myocardial Infarction; Acute Coronary Syndrome; Metabolic Disturbance
Keywords: Myocardial Infarction; Acute Coronary Syndrome; Standard modifiable risk factor; Metabolomic biomarkers
MeSH Terms: conditions — Cardiovascular Diseases; Acute Coronary Syndrome; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Centrifuged blood chemistry test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SMuRFs: Patients with acute myocardial infraction with a history of at least one standard modifiable risk factor (SMuRF; smoking, diabetes mellitus, dyslipidemia, hypertension)
  Interventions: Diagnostic Test: Investigation of the metabolic substrate
- SMuRF-less: Patients with acute myocardial infraction without history of any SMuRF
  Interventions: Diagnostic Test: Investigation of the metabolic substrate

INTERVENTIONS:
Diagnostic Test: Investigation of the metabolic substrate — A blood sample will be received from each patient to assess novel metabolomic biomarkers' levels at the time of acute myocardial infraction

SUMMARY:
Coronary heart disease (CHD) is the leading cause of mortality worldwide. Every year, millions of people suffer its most adverse manifestation, an acute myocardial infraction (AMI). The majority of these patients present at least one of the standard modifiable risk factors (SMuRFs). These include smoking, hypertension, dyslipidemia, and diabetes mellitus (DM). However, emerging scientific evidence recognizes a clinically significant proportion of patients presenting with life-threatening AMI without any SMuRF (SMuRF-less patients). This proportion of patients with ACS without SMuRF appears to be increasing during the last two decades and has recently been reported as high as 20% (of total AMIs). To date, there are no scientific data capable of highlighting specific risk factors-biomarkers responsible for the development of AMIs SMuRF-less patients. Concurrently, metabolomics is rapidly evolving as a novel technique of studying small molecule substrates, intermediates and products of cell metabolism. This technique could be utilized to flag patients with higher risk for increased atherosclerotic burden, and subsequent future adverse clinical events. Besides the already established biomarkers, several metabolomic indicators, such as ceramides (C16, C18 και C24), acylcarnitines, apolipoproteins (ApoΒ and ApoA1) and adiponectin, have been separately shown to increase the risk for coronary artery disease development and progression. Therefore, the two groups of patients (with SMuRFs vs SMuRF-less) will be compared regarding their metabolic fingerprints -specifically the aforementioned novel metabolomic biomarkers- and possible predictive factors leading to SMuRF-less AMI will be evaluated. On the basis of the above, the aim is to prospectively analyze a cohort of well-characterized patients with AMI. The rationale of the study is to investigate potential correlations between metabolic profile of patients and SMuRF-less AMI. This could lead to the development of predictive risk stratification algorithms for patients without SMuRFs and coronary artery disease.

DETAILED DESCRIPTION:
Coronary heart disease (CHD) is the leading cause of mortality worldwide. Every year, millions of people suffer its most adverse manifestation, an acute myocardial infraction (AMI). The majority of these patients present at least one of the standard modifiable risk factors (SMuRFs). These include smoking, hypertension, dyslipidemia, and diabetes mellitus (DM). However, emerging scientific evidence recognizes a clinically significant proportion of patients presenting with life-threatening AMI without any SMuRF (SMuRF-less patients). This proportion of patients with ACS without SMuRF appears to be increasing during the last two decades and has recently been reported as high as 20% (of total AMIs). To date, there are no scientific data capable of highlighting specific risk factors-biomarkers responsible for the development of AMIs SMuRF-less patients.

Concurrently, metabolomics is rapidly evolving as a novel technique of studying small molecule substrates, intermediates and products of cell metabolism. This technique could be utilized to flag patients with higher risk for increased atherosclerotic burden, and subsequent future adverse clinical events. Besides the already established biomarkers, several metabolomic indicators, such as ceramides (C16, C18 και C24), acylcarnitines, apolipoproteins (ApoΒ and ApoA1) and adiponectin, have been separately shown to increase the risk for coronary artery disease development and progression. Therefore, the two groups of patients (with SMuRFs vs SMuRF-less) will be compared regarding their metabolic fingerprints -specifically the aforementioned novel metabolomic biomarkers- and possible predictive factors leading to SMuRF-less AMI will be evaluated. On the basis of the above, the aim is to prospectively analyze a cohort of well-characterized patients with AMI. The rationale of the study is to investigate potential correlations between metabolic profile of patients and SMuRF-less AMI. This could lead to the development of predictive risk stratification algorithms for patients without SMuRFs and coronary artery disease.

Blood tests (blood chemistry) will be received from each patient on admission and will be analyzed to assess patients' metabolic profile. In order to achieve full coverage of all compounds, different analytical platforms and methods, such as Enzyme-LInked Immunosorbent Assay (ELISA), Reversed Phase Liquid Chromatography tandem Mass Spectrometry (RPLC-MS/MS) and Hydrophilic Interaction Liquid Chromatography tandem Mass Spectrometry (HILIC-MS/MS) will be applied. Univariate and multivariate analysis with linear and logistic regression models will be used to investigate independent prognostic factors contributing to the occurrence of SMuRF-less AMIs. The potential application in daily clinical practice of a derived clinical predictive model-algorithm, possibly including a new panel of metabolomic biomarkers, will contribute to the early prognosis and personalized prevention of such a particular category of AMIs.

ELIGIBILITY:
Inclusion Criteria:

* Age >25 years
* Hospitalization for acute myocardial infarction (AMI) with or without ST elevation (based on Fourth Universal Definition of Myocardial Infarction) within the previous 4 weeks
* Coronary angiography before or after hospitalization for AMI, in which at least one stenosis >50% in a major epicardial coronary artery (left anterior descending artery, left circumflex artery, right coronary artery) or a branch thereof with a diameter of at least 2 mm was observed.

Exclusion Criteria:

* Inability or refusal to provide informed consent
* Age >80 years
* History of hospitalization due to AMI prior to the present AMI
* History of coronary revascularization prior to the present AMI AMI
* Previous coronary angiography (prior to the present AMI) showing >50% stenosis in a major epicardial coronary artery

Exclusion Criteria for SMuRF-less patients group only:

* Known history of hypertension and/or antihypertensive treatment prior to AMI
* Use of tobacco products on a systematic basis for up to <12 months before AMI
* History of diabetes mellitus type 1 or 2 and/or treatment with antidiabetic tablets or insulin before AMI or diagnosis of diabetes mellitus based on HbA1c during AMI hospitalization
* Known hypercholesterolemia (total chol >200 mg/dl / LDLc >150 mg/dl) or treatment with statins or PCSK9is, before AMI

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients >25years old presenting with acute myocardial infraction with or without ST elevation within the previous 4 weeks, with at least one angiographically-testified stenosis>50% in a major epicardial coronary artery
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-10-15 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Metabolomic biomarkers associated with SMuRF-less myocardial infraction | 3 years
  Identification of differences in metabolomic biomarkers' levels (metabolic substrate) between SMuRF-less myocardial infractions and myocardial infractions in patients with SMuRFs

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Moysidis, Study Chair — Aristotle University Of Thessaloniki